CLINICAL TRIAL: NCT07274670
Title: A Randomized Double-Blind Controlled Trial on the Effectiveness of Superficial Cervical Plexus Block With Dexmedetomidine Compared to Without Adjuvant in Thyroid Surgery
Brief Title: Superficial Cervical Plexus Block With Dexmedetomidine Versus Without Adjuvant in Thyroid Surgery
Acronym: BPSS-DEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Lya Lusyana, Anesthesiology and Intensive Therapy Specialist Program Resident Doctor, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYA-BPSS-DEX-2025; Institutional Review Board (Other: No : 1805/UN14.2.2.VII.14/LT/2025)
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Cancer; Goiter; Hyperthyroidism
Keywords: Superficial Cervical Plexus Block; SCPB; Dexmedetomidine; Thyroidectomy; Postoperative Pain; Chronic Pain
MeSH Terms: conditions — Thyroid Neoplasms; Goiter; Hyperthyroidism; Pain, Postoperative; Chronic Pain | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel arms with a 1:1 allocation ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study. The following measures ensure blinding:
  Intervention Blinding: The preparation and mixing of the local anesthetic solution (with or without Dexmedetomidine adjuvant) are performed by a third party not involved in the execution of the block or patient follow-up. The final solutions are made to look identical.
  Investigator/Assessor Blinding: The principal investigator and the Acute Pain Service (APS) team that performs post-operative assessments (VAS scores, opioid consumption, complications, and long-term follow-up) are blinded to the treatment group allocation (Dexmedetomidine or control).
  Participant Blinding: Participants are informed that the difference lies only in the adjuvant given, thus they are blinded to the specific substance received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCPB with Dexmedetomidine Adjuvant (Experimental): Patients receive Superficial Cervical Plexus Block (SCPB) with Bupivacaine 0.375% and Dexmedetomidine 0.5 mcg/kgbw
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- SCPB with Placebo/No Adjuvant (Active Comparator): Patients receive Superficial Cervical Plexus Block (SCPB) with Bupivacaine 0.375% only (without Dexmedetomidine adjuvant).
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine & Bupivacaine. — Superficial Cervical Plexus Block (SCPB) performed under ultrasound guidance (in-plane technique). The regimen consists of Bupivacaine 0.375% with the adjuvant Dexmedetomidine at a dose of 0.5 mcg/kgbw. The total volume injected is 20 mL (10 mL on each side) into the fascial space between the sternocleidomastoid muscle and the prevertebral fascia. The block is performed after induction of general anesthesia
  Other Names: Dexmedetomidine; Bupivacaine; BPSS
  Arms: SCPB with Dexmedetomidine Adjuvant
Drug: Bupivacain — Superficial Cervical Plexus Block (SCPB) performed under ultrasound guidance (in-plane technique). The regimen consists of Bupivacaine 0.375% only. The total volume injected is 20 mL (10 mL on each side) [cite_start], supplemented with Saline/Placebo to match the volume and appearance of the active drug. The block is performed after induction of general anesthesia.
  Other Names: Bupivacaine; BPSS
  Arms: SCPB with Placebo/No Adjuvant

SUMMARY:
Efficacy of Superficial Cervical Plexus Block (SCPB) with Dexmedetomidine Adjuvant Compared to Without Adjuvant in Thyroid Surgery. This is a double-blinded, randomized controlled trial designed to evaluate the effectiveness of adding perineural dexmedetomidine to a Superficial Cervical Plexus Block (SCPB) for pain management in patients undergoing thyroid surgery. The study aims to prove that SCPB with dexmedetomidine adjuvant provides superior post-operative analgesia, lowers total opioid consumption, prolongs the time until the first analgesic request, and reduces the incidence of chronic pain three months post-surgery compared to SCPB without the adjuvant. The study will also evaluate the anti-inflammatory effect by measuring the reduction in Interleukin-6 (IL-6) levels post-operatively and compare the incidence of bradycardia as a side effect. The total required sample size is 58 subjects.

DETAILED DESCRIPTION:
Thyroid surgery is a major procedure often associated with acute and chronic postoperative pain in the neck area. Chronic post-surgical pain can significantly affect the patient's long-term quality of life. Superficial Cervical Plexus Block (SCPB) is an effective regional anesthesia technique used to manage perioperative pain and reduce the need for postoperative opioids. However, achieving an optimal duration of analgesia remains a challenge. Dexmedetomidine, an alpha_2-adrenergic receptor agonist, is frequently used as an adjuvant to prolong the analgesic effect of nerve blocks. Studies have shown that combining dexmedetomidine with SCPB provides better and longer-lasting analgesia. Dexmedetomidine also possesses anti-inflammatory properties, potentially lowering the level of Interleukin-6 (IL-6), a biomarker of inflammation often elevated after surgery that can exacerbate pain. The effectiveness of SCPB with dexmedetomidine adjuvant, particularly in reducing inflammation and chronic pain incidence, has not been widely explored locally at RSUP Prof. Dr. I.G.N.G. Ngoerah.Study Objectives: The primary goal is to prove the effectiveness of dexmedetomidine as an SCPB adjuvant in thyroid surgery, assessed by acute and chronic pain outcomes. Acute Pain Outcomes: Measured by Visual Analogue Scale (VAS) scores at 6, 12, and 24 hours post-operation, time to first Patient-Controlled Analgesia (PCA) button press, total opioid consumption via PCA over 24 hours, and changes in the inflammatory biomarker Interleukin-6 (IL-6). Chronic Pain Outcomes: Measured by the incidence of chronic pain three months post-surgery using the Brief Pain Inventory Short Form (BPI-SF) questionnaire. Safety Outcome: Measured by the incidence of bradycardia. Correlations: To prove the correlation between the change in Interleukin-6 levels with 24-hour pain scores and the incidence of chronic pain.Study Design and Intervention: This is a true experimental study with a double-blinded randomized pre- and post-control group design. Group P1 (Intervention): Patients receive SCPB with 0.375% Bupivacaine plus 0.5 mcg/kgbw Dexmedetomidine (total volume 20 mL, injected 10 mL on each side). Group P2 (Control): Patients receive SCPB with 0.375% Bupivacaine only (total volume 20 mL, injected 10 mL on each side).All procedures are performed under general anesthesia with Ultrasound guidance. Analgesia management includes PCA Fentanyl and combination analgesics (Paracetamol and Ibuprofen). The minimum required sample size is 58 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-59 years.
* Patients with ASA physical status classification I-III.
* Patients with Body Mass Index (BMI) between 18 and 25 kg/m

Exclusion Criteria:

* Patients with contraindications for regional anesthesia.
* Patients with a history of autoimmune disease.
* Presence of infection in the puncture area.
* Patients with allergies and contraindications to the use of dexmedetomidine.
* Patients on routine medication, including beta-blockers, anti-depressants, or anti-seizure medications.
* Prolonged opioid use.
* Patients unable to be assessed using the Visual Analogue Scale (VAS) or unable to operate the Patient-Controlled Analgesia (PCA) device.
* Patients who refuse to participate in the study.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Time to First Request for Opioid Analgesia (PCA Button Press) | up to 24 hours post-operation ( 1440 minutes )
  From the time of PCA activation in the Post-Anesthesia Care Unit (PACU) until the completion of the first 24 hours post-operation. The cumulative consumption of Fentanyl (in micrograms) is recorded from the PCA device's counter, with the assessment period duration calculated precisely in minutes

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score at 6, 12, and 24 Hours Post-Operation | 6 hours, 12 hours, and 24 hours post-operation.
  Assessment of acute pain intensity using the Visual Analogue Scale (VAS) (0-100 mm, where 0 is no pain and 100 is the worst pain imaginable).
Total Fentanyl Opioid Consumption in the First 24 Hours Post-Operation | 24 hours post-operation
  The total amount of fentanyl (in mcg) consumed by the patient via the Patient-Controlled Analgesia (PCA) device.
Change in Interleukin-6 (IL-6) Level Post-Operation | Measured as the difference between 24 hours post-operation and pre-general anesthesia.
  The delta change ($\Delta$) in plasma Interleukin-6 (IL-6) concentration (in pg/mL) comparing the pre-operative baseline to the 24-hour post-operative measurement.
Incidence of Chronic Pain at 3 Months Post-Operation | 3 months post-operation (90 days)
  Incidence of Chronic Post-Surgical Pain (CPSP) defined by the Brief Pain Inventory Short Form (BPI-SF) score (any score > 0) lasting longer than three months.

CONTACTS AND LOCATIONS:
Overall Officials: Lya Lusyana, dr., Study Chair — Universitas Udayana; Pontisomaya Parami, Sp.An, Study Director — Universitas Udayana; I Gusti Ngurah Mahaalit Arimbawa, Sp.An, Study Director — Universitas Udayana
Locations (1):
- Prof. Dr. I.G.N.G Ngoerah Central General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Udayana University Official Website — https://www.unud.ac.id/